CLINICAL TRIAL: NCT01997593
Title: Evaluate the Analgesic Effect of Intraperitoneal Infiltration of Ropivacaine in Children Undergoing Laparoscopic Surgery
Brief Title: Peritoneal Ropivacaine Infiltration on Postoperative Pain in Children Affected
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ping Yang (Other)
Responsible Party: Sponsor-Investigator, Ping Yang, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 20130801
Record Dates: First submitted 2013-10-27; First posted 2013-11-28 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Testicular; Colic
Keywords: analgesia; pediatric; pain; laparoscopy; ropivacaine
MeSH Terms: conditions — Colic; Agnosia; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- ropivacaine (Experimental): Preincisional wound intraperitoneal infiltration of 1% ropivacaine 0.3ml/kg was performed in group I patients before surgery.
  Interventions: Drug: intraperitoneal infiltration of ropivacaine

INTERVENTIONS:
Drug: intraperitoneal infiltration of ropivacaine — intraperitoneal infiltration of ropivacaine by a special equipment

SUMMARY:
The aim of this study was to evaluate the analgesic effect of intraperitoneal infiltration of ropivacaine in children undergoing laparoscopic surgery.

DETAILED DESCRIPTION:
1. Quality assurance plan that addresses data validation and registry procedures, including any plans for site monitoring and auditing.
2. Data checks to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.
3. Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources .
4. Data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, coding information .
5. Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management.
6. Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect.
7. Plan for missing data to address situations where variables are reported as missing, unavailable, "non-reported," uninterpretable, or considered missing because of data inconsistency or out-of-range results
8. Statistical analysis plan describing the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives, as specified in the study protocol or plan

ELIGIBILITY:
Inclusion Criteria:

1. Between 6 months and 5years.
2. Laparoscopic inguinal hernia repair
3. Laparoscopic testicular descent fixation

Exclusion Criteria:

1. Patient who are suffering from mental disease
2. Patient who suffering from neuromuscular disease
3. Local anesthetic allergy
4. Patient who needs directly into ICU after the operation.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
pain score | within the first 2days after the surgery

SECONDARY OUTCOMES:
Analgesic dose | Within the first 2days after the surgery
Gastrointestinal function recovery score | Within the first 2days after the surgery
Wound score | Within the first 2days after the surgery
Time to discharge | Participants will be followed for the duration of hospital stay, an expected average of 2weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yang Hui, Professor, Study Director — China Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China